CLINICAL TRIAL: NCT06947096
Title: A Prospective Clinical Study of Radiomics-Based Artificial Intelligence for Predicting Para-Aortic Lymph Node Metastasis in Patients With Gastric Cancer
Brief Title: Radiomics-Based AI Model for Predicting Para-Aortic Lymph Node Metastasis in Gastric Cancer Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Qun Zhao (Other)
Collaborators: First Hospital of Shijiazhuang City (Other); Baoding First Central Hospital (Other); Hengshui People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Qun Zhao, Professor, Hebei Medical University
Organization: Hebei Medical University (Other)
Other Study IDs: GC-RAD-AI-2025-01
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Gastric Cancer; Para-Aortic Lymph Node Metastasis; Lymphatic Metastasis; Preoperative Imaging Assessment; Radiomics; Artificial Intelligence
MeSH Terms: conditions — Stomach Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Radiomics-Based AI Imaging Analysis — This intervention involves the development and application of a radiomics-based artificial intelligence (AI) model to analyze preoperative abdominal CT images of patients with gastric cancer. The AI algorithm extracts high-dimensional imaging features from the para-aortic region to predict the presence or absence of para-aortic lymph node metastasis (PALNM). This non-invasive method aims to assist clinicians in preoperative risk stratification and treatment planning. The model will be trained and validated using manually segmented lymph node regions and correlated with postoperative pathological findings to ensure accuracy and clinical relevance.

SUMMARY:
This study aims to develop and validate an artificial intelligence (AI) model based on radiomics features extracted from preoperative CT images to predict para-aortic lymph node (PALN) metastasis in patients with gastric cancer. Accurately identifying PALN metastasis before surgery can help doctors make better treatment decisions, such as whether to proceed with surgery, consider chemotherapy, or use other treatment strategies. The study will prospectively enroll patients who are diagnosed with gastric cancer and scheduled for surgery. All participants will undergo routine imaging tests, and their data will be analyzed using advanced AI techniques. The results of this study may improve the precision of preoperative staging and support personalized treatment planning for gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-80 years.
2. Histologically confirmed gastric adenocarcinoma.
3. Planned to undergo radical gastrectomy with or without para-aortic lymph node dissection.
4. Preoperative contrast-enhanced abdominal CT scan available within 3 weeks before surgery.
5. No evidence of distant metastasis on imaging.
6. ECOG performance status 0-2.
7. Provided written informed consent.

Exclusion Criteria:

1. History of other malignant tumors within the past 5 years.
2. Received neoadjuvant chemotherapy or radiotherapy prior to CT imaging.
3. Poor-quality or incomplete CT images not suitable for radiomics analysis.
4. Severe comorbidities that may affect prognosis or surgical decision-making.
5. Pregnancy or breastfeeding.
6. Inability to provide informed consent or comply with study procedures.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients diagnosed with gastric adenocarcinoma who are scheduled to undergo radical gastrectomy at a tertiary care center. All participants will have preoperative contrast-enhanced CT scans and no evidence of distant metastasis. The population represents individuals at risk of para-aortic lymph node metastasis, and is intended to reflect real-world patients who may benefit from non-invasive, AI-assisted preoperative assessment tools. Participants will be enrolled consecutively to minimize selection bias.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of the AI Radiomics Model for Predicting Para-Aortic Lymph Node Metastasis in Gastric Cancer | From Preoperative Imaging to Postoperative Pathological Confirmation (Approximately 4-6 Weeks per Patient)
  The primary outcome is the diagnostic performance of the radiomics-based AI model in predicting para-aortic lymph node metastasis (PALNM) in patients with gastric cancer. Performance will be evaluated by calculating the area under the receiver operating characteristic curve (AUC), sensitivity, specificity, accuracy, and predictive values. The ground truth for PALNM status will be based on postoperative pathological findings or multidisciplinary consensus diagnosis. The model's predictions will be compared with actual clinical outcomes to assess its reliability and clinical utility.

CONTACTS AND LOCATIONS:
Locations (1):
- the Fourth Hospital of Hebei Medical University, Shijiazhuang, None Selected, China